CLINICAL TRIAL: NCT01808248
Title: A Phase 2, Open-Label Study of Sofosbuvir in Combination With PEG and Ribavirin for 12 Weeks in Treatment Experienced Subjects With Chronic HCV Infection Genotype 2 or 3
Brief Title: Sofosbuvir (GS-7977) in Combination With PEG and Ribavirin for 12 Weeks in Treatment Experienced Subjects With Chronic HCV Infection Genotype 2 or 3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-334-0151
Expanded Access: NCT01779518 (Approved for marketing)
Record Dates: First submitted 2013-03-01; First posted 2013-03-11 (Estimated); Results first posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Hepatitis C
Keywords: HCV genotype 2 (GT-2); HCV genotype 3 (GT-3); HCV; Sustained Virologic Response; Direct Acting Antiviral; Combination Therapy; Treatment-Naïve; GS-7977; Ribavirin; RBV; Peginterferon Alfa 2a; PEG; Additional relevant MeSH terms:; Hepatitis; Hepatitis A; Hepatitis, Chronic; Hepatitis C; Hepatitis C, Chronic; Liver Diseases; Digestive System Diseases; Hepatitis, Viral, Human; Virus Diseases; Enterovirus Infections; Picornaviridae Infections; RNA Virus Infections; Flaviviridae Infections; Peginterferon alfa-2a; Interferon-alpha; Antiviral Agents; Anti-Infective Agents; Therapeutic Uses; Pharmacologic Actions; Antimetabolites; Molecular Mechanisms of Pharmacological Action; Immunologic Factors; Physiological Effects of Drugs
MeSH Terms: conditions — Hepatitis C; Hepatitis; Hepatitis A; Hepatitis, Chronic; Hepatitis C, Chronic; Liver Diseases; Digestive System Diseases; Hepatitis, Viral, Human; Virus Diseases; Enterovirus Infections; Picornaviridae Infections; RNA Virus Infections; Flaviviridae Infections | interventions — Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SOF+PEG+RBV (Experimental): Participants will receive SOF+PEG+RBV for 12 weeks.
  Interventions: Drug: SOF; Drug: PEG; Drug: RBV

INTERVENTIONS:
Drug: SOF — Sofosbuvir (SOF) 400 mg tablet administered orally once daily
  Other Names: Sovaldi®; GS-7977; PSI-7977
Drug: PEG — Peginterferon alfa 2a (PEG) 180 μg administered once weekly by subcutaneous injection
Drug: RBV — Ribavirin (RBV) tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75kg = 1000 mg and ≥ 75 kg = 1200 mg)

SUMMARY:
This study is to evaluate the safety, tolerability, and antiviral efficacy of sofosbuvir (SOF) in combination with peginterferon alfa 2a (PEG) and ribavirin (RBV) administered for 12 weeks in participants with chronic genotype 2 or 3 hepatitis C virus (HCV) infection who have previously failed prior treatment with an interferon-based regimen.

ELIGIBILITY:
Inclusion Criteria:

* Infection with genotype 2 or 3 HCV infection
* Cirrhosis determination
* Individual is treatment-experienced
* Screening laboratory values within defined thresholds
* Individual has not been treated with any investigational drug or device within 30 days of the Screening visit
* Use of highly effective contraception methods if female of childbearing potential or sexually active male

Exclusion Criteria:

* Prior exposure to a direct-acting antiviral drug targeting the HCV NS5B polymerase
* Pregnant or nursing female or male with pregnant female partner
* Current or prior history of clinical hepatic decompensation
* History of clinically-significant illness or any other major medical disorder that may interfere with treatment, assessment, or compliance with the study protocol
* Excessive alcohol ingestion or significant drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-02; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rob Hyland, Study Director — Gilead Sciences
Locations (1):
- Alamo Medical Research, San Antonio, Texas, United States

REFERENCES:
- See also: Medicine Plus — http://www.nlm.nih.gov/medlineplus/
- See also: Hepatitis — http://www.nlm.nih.gov/medlineplus/hepatitis.html
- See also: Hepatitis A — http://www.nlm.nih.gov/medlineplus/hepatitisa.html
- See also: Hepatitis C — http://www.nlm.nih.gov/medlineplus/hepatitisc.html
- See also: Drug Information available for: — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp
- See also: Ribavirin — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=0036791045&QV1=RIBAVIRIN
- See also: PEGINTERFERON ALFA-2A — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=0198153514&QV1=PEGINTERFERON+ALFA-2A
- See also: U.S. FDA Resources — http://clinicaltrials.gov/ct2/info/fdalinks

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a single site in the United States. The first participant was screened on 18 February 2013. The last participant observation occurred on 06 December 2013.
Pre-assignment Details: 56 participants were screened; 47 participants were enrolled and treated, and comprise the Safety Analysis Set and the Full Analysis Set.
Groups:
- SOF+PEG+RBV: Sofosbuvir (SOF) 400 mg tablet once daily + peginterferon alfa 2a (PEG) 180 μg subcutaneous injection once weekly + weight-based ribavirin (RBV; 1000-1200 mg as 200 mg tablets in a divided daily dose) for 12 weeks.
Period: Overall Study
Arm/Group | SOF+PEG+RBV
Started | 47
Completed Posttreatment Week 12 Visit | 45
Completed | 42
Not Completed | 5
Not completed — Lack of Efficacy | 3
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants enrolled and received at least 1 dose of study drug
Groups:
- Genotype 2: SOF 400 mg tablet once daily + PEG 180 μg subcutaneous injection once weekly + weight-based RBV (1000-1200 mg as 200 mg tablets in a divided daily dose) for 12 weeks in participants with genotype 2 hepatitis C virus (HCV) infection.
- Genotype 3: SOF 400 mg tablet once daily + PEG 180 μg subcutaneous injection once weekly + weight-based RBV (1000-1200 mg as 200 mg tablets in a divided daily dose) for 12 weeks in participants with genotype 3 HCV infection.
- Total: Total of all reporting groups
Arm/Group | Genotype 2 | Genotype 3 | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (6.1) | 54 (6.9) | 56 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 14 | 18 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 10 | 21
  Not Hispanic or Latino | 12 | 14 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 0 | 1 | 1
  White | 22 | 23 | 45
  Asian | 1 | 0 | 1
Liver Cirrhosis [Number; unit: participants]
  No | 9 | 12 | 21
  Yes | 14 | 12 | 26
IL28b Status [Number; unit: participants] — CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 10 | 7 | 17
    CT | 10 | 15 | 25
    TT | 3 | 2 | 5
HCV RNA (log10 IU/mL) [Mean (Standard Deviation); unit: log10 IU/mL] | 6.4 (0.66) | 6.0 (0.62) | 6.2 (0.66)
HCV RNA Category [Number; unit: participants]
  < 6 log10 IU/mL | 4 | 13 | 17
  ≥ 6 log10 IU/mL | 19 | 11 | 30
Response to prior HCV treatment [Number; unit: participants]
  Nonresponse | 2 | 5 | 7
  Relapse/Breakthrough | 21 | 19 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) at 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, < 15 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants with genotype 2 or 3 HCV infection who were enrolled and received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Groups:
- Genotype 2: SOF 400 mg tablet once daily + PEG 180 μg subcutaneous injection once weekly + weight-based RBV (1000-1200 mg as 200 mg tablets in a divided daily dose) for 12 weeks in participants with genotype 2 HCV infection.
Arm/Group | Genotype 2 | Genotype 3
Number analyzed (Participants) | 23 | 24
percentage of participants | 95.7 | 83.3

2. Primary Outcome: Incidence of Adverse Events Leading to Permanent Discontinuation of Study Drug(s)
Description: The percentage of participants discontinuing any study drug due to an adverse event was summarized.
Time Frame: Up to 12 weeks
Population: Safety Analysis Set: participants enrolled and received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Groups:
- SOF+PEG+RBV: SOF 400 mg tablet once daily + PEG 180 μg subcutaneous injection once weekly + weight-based RBV (1000-1200 mg as 200 mg tablets in a divided daily dose) for 12 weeks.
Arm/Group | SOF+PEG+RBV
Number analyzed (Participants) | 47
percentage of participants | 8.5

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response at 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR24 were defined as HCV RNA < LLOQ at 4 and 24 weeks following the last dose of study drug, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Genotype 2 | Genotype 3
Number analyzed (Participants) | 23 | 24
percentage of participants
  SVR4 | 95.7 | 87.5
  SVR24 | 95.7 | 83.3

4. Secondary Outcome: Percentage of Participants Experiencing On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as:
  1. Viral breakthrough: HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment, confirmed with 2 consecutive values (second confirmation value may have been posttreatment) or with a last available on-treatment measurement and no subsequent follow-up values, or
  2. Viral rebound: > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment, confirmed with 2 consecutive values (second confirmation value may have been posttreatment) or with a last available on-treatment measurement and no subsequent follow-up values, or
  3. Nonresponse: HCV RNA persistently ≥ LLOQ through 8 weeks of treatment
Time Frame: Up to 12 weeks
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Genotype 2 | Genotype 3
Number analyzed (Participants) | 23 | 24
percentage of participants | 0 | 0

5. Secondary Outcome: Percentage of Participants Experiencing Viral Relapse
Description: Viral relapse was defined as having HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at the end of treatment, confirmed with 2 consecutive values or last available posttreatment measurement.
Time Frame: Up to Posttreatment Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Genotype 2 | Genotype 3
Number analyzed (Participants) | 22 | 23
percentage of participants | 0 | 8.7

ADVERSE EVENTS:
Time Frame: Up to 12 weeks plus 30 days
Arm/Group | SOF+PEG+RBV
Serious Adverse Events (participants affected / at risk) | 4/47
Other Adverse Events (participants affected / at risk) | 45/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+PEG+RBV (N=47)
Anaemia (Blood and lymphatic system disorders) | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Sepsis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+PEG+RBV (N=47)
Anaemia (Blood and lymphatic system disorders) | 14
Neutropenia (Blood and lymphatic system disorders) | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 7
Nausea (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 5
Aphthous stomatitis (Gastrointestinal disorders) | 3
Influenza like illness (General disorders) | 26
Fatigue (General disorders) | 15
Upper respiratory tract infection (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 3
Decreased appetitie (Metabolism and nutrition disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 7
Dizziness (Nervous system disorders) | 4
Insomnia (Psychiatric disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 7
Pruritis (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years